CLINICAL TRIAL: NCT02191917
Title: A Study of Respiratory Muscle Strength, Including Effort-Independent Measures, in Subjects With Late-Onset Pompe Disease
Brief Title: A Study of Respiratory Muscle Strength in Patients With Late-onset Pompe Disease (LOPD)
Status: Terminated | Type: Observational
Why Stopped: Study was terminated early due to a company decision not based on safety concerns
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 701-201; 2014-002158-38 (EudraCT Number)
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Results first posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-04

CONDITIONS: Late-onset Pompe Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Measurement of Respiratory Muscle Strength
  Interventions: Procedure: Respiratory muscle strength measurements by different techniques.

INTERVENTIONS:
Procedure: Respiratory muscle strength measurements by different techniques.

SUMMARY:
Study 701-201 is a study in patients with late-onset Pompe disease (LOPD). The study will test respiratory muscle strength initially and again after 24 weeks in subjects treated or not treated with BMN 701 .

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent, after the nature of the study has been explained, and prior to any study-related procedures
* Documented diagnosis with late-onset Pompe disease - At least 18 years of age at study entry
* Willing and able to comply with all study procedures

Exclusion Criteria:

* Requires ventilatory support while awake and in the upright position
* Concurrent disease, medical condition, or extenuating circumstance that, in the opinion of the investigator, might compromise patient well-being, study completion, or data collection
* Allergy to tools or procedures used for respiratory muscle testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifteen subjects were planned for enrollment; there were no screening failures; 8 subjects were enrolled. Two subjects were enrolled from 701-301 and the remaining 6 subjects enrolled directly into 701-201 (no parent study)
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-10-21 (Actual); Primary Completion 2016-06-22 (Actual); Study Completion 2016-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — BioMarin Pharmaceutical
Locations (2):
- University of Florida, Gainesville, Florida, United States
- Royal Brompton Hospital, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall: All enrolled subjects
Period: Overall Study
Arm/Group | Overall
Started | 8
Completed | 7
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall: All subjects
Arm/Group | Overall
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  Other | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 7
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximal Inspiratory Pressure (MIP)
Description: Pulmonary measure of change in maximal inspiratory pressure (MIP)
Time Frame: Baseline, Week 28
Population: Full Analysis Set (FAS) population includes all enrolled subjects who have at least one study assessment.
Measure: Mean (Standard Deviation); unit: cm H2O
Groups:
- Overall: All participants
Arm/Group | Overall
Number analyzed (Participants) | 8
cm H2O
  Baseline | 49.2 (21.7)
  Last Visit: number analyzed (Participants) | 7
  Last Visit | 46.0 (20.93)
  Change from Baseline: number analyzed (Participants) | 7
  Change from Baseline | -5.5 (8.38)

2. Secondary Outcome: Maximal Expiratory Pressure (MEP)
Description: Pulmonary measure of change in maximal expiratory pressure (MEP)
Time Frame: Baseline, Week 28
Population: Full Analysis Set (FAS) population includes all enrolled subjects who have at least one study assessment.
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Overall
Number analyzed (Participants) | 8
cm H2O
  Baseline | 77.1 (32.39)
  Last Visit: number analyzed (Participants) | 7
  Last Visit | 69.0 (24.18)
  Change from Baseline: number analyzed (Participants) | 7
  Change from Baseline | -11.6 (11.35)

ADVERSE EVENTS:
Time Frame: 28 weeks
Groups:
- Overall: Overall
Arm/Group | Overall
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=8)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was planned to have 15 participants. However, the study was terminated prematurely. Only 8 participants were enrolled. Seven participants had last assessment at Days 146, 168, 172, 174, 179, 188, 196, translating to one participant at Week 20 and six participants Weeks 24-28.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days